CLINICAL TRIAL: NCT07388095
Title: Neoadjuvant Treatment With Adebrelimab in Combination With Nimotuzumab and Chemotherapy for Resectable Esophageal Squamous Cell Carcinoma: A Single-arm, Exploratory Phase II Clinical Study
Brief Title: Adebrelimab Neoadjuvant Treatment for Resectable ESCC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: neoESCC-001
Record Dates: First submitted 2026-01-23; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: ESCC
MeSH Terms: interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Adebrelimab+Nimotuzumab+chemotherapy
  Interventions: Drug: Adebrelimab (PD-L1 inhibitor)

INTERVENTIONS:
Drug: Adebrelimab (PD-L1 inhibitor) — Adebrelimab: 1200mg, iv, d1, Q3W, 2cycles Nimotuzumab:400 mg, d1,d8, Q3W, 2cycles Cisplatin: 75mg/m2，d1, Q3W, 2cycles Albumin-bound paclitaxel: 260 mg/m2, d1, Q3W, 2cycles

SUMMARY:
This is a prospective, phase II, exploratory clinical trial.

The study aims to evaluate the efficacy and safety of in combination adebrelimab with nimotuzumab and chemotherapy as neoadjuvant therapy in patients with resectable esophageal squamous cell carcinoma.

The primary endpoint is pCR ( pathological complete response), evaluating the efficacy of adebrelimab in combination with nimotuzumab and neoadjuvant chemotherapy in patients with resectable esophageal squamous cell carcinoma. After the primary objective is achieved, EFS (event free survival ), R0 resection rate, MPR (major pathological response), OS (overall survival), and safety will be assessed as key secondary objectives. The study plans to enroll 22 patients with resectable esophageal squamous cell carcinoma.

The study is divided into a screening period, a treatment period, and a follow-up period. Subjects will enter the screening period after signing informed consent. Subjects who pass the screening assessment will be enrolled in the study. Eligible subjects will receive two cycles of neoadjuvant therapy with adebrelimab, nimotuzumab, nab-paclitaxel, and cisplatin. Esophagectomy will be performed after two cycles of neoadjuvant therapy (4-6 weeks after the last dose). Researchers will determine subsequent treatment based on postoperative pathology. After treatment (surgery), safety and efficacy follow-ups will commence. When a subject first experiences disease progression as assessed by the investigator according to RECIST v1.1, confirmation is required after 4-6 weeks (except for rapid or significant clinical progression). Subjects whose disease progression is not confirmed by imaging after 4-6 weeks may continue treatment if their clinical symptoms remain stable, as determined by the investigator, until imaging-confirmed disease progression occurs, or other termination criteria as specified in the protocol are met, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent to voluntarily participate in this study;
2. Pathologically confirmed resectable esophageal squamous cell carcinoma (excluding mixed adenocarcinoma-squamous cell carcinoma types);
3. Thoracic esophageal cancer confirmed by CT/MRI/EUS assessment with clinical stage IIA-IIIB (according to AJCC 8th edition);
4. Age 18-75 years, male or female;
5. ECOG PS 0-1;
6. No prior anticancer treatment for esophageal cancer, including radiotherapy, chemotherapy, or surgery;
7. Planned surgical treatment following completion of neoadjuvant therapy;
8. No surgical contraindications;
9. Normal major organ function, including: (1) Complete blood count (no use of blood components, cell growth factors, leukocyte-stimulating agents, platelet-stimulating agents, or anemia-correcting agents within 14 days prior to first study drug administration): White blood cell count ≥ 4.0 × 10^9/L Neutrophil count ≥ 1.5 × 10^9/L Platelet count ≥ 90 × 10^9/L Hemoglobin ≥ 90 g/L (2) Blood Biochemistry Tests: Total Bilirubin ≤ 1.5×ULN, LT ≤ 2.5×ULN, AST ≤ 2.5×ULN, Serum Creatinine ≤ 1.5×ULN, or Creatinine Clearance ≥ 50 mL/min (Cockcroft-Gault formula) c) Coagulation Function: International Normalized Ratio (INR) ≤ 1.5×ULN Activated Partial Thromboplastin Time (APTT) ≤ 1.5×ULN
10. Female subjects of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to initiation of study drug administration and must use effective contraception (e.g., intrauterine device, oral contraceptives, or condoms) during the trial and for at least 3 months after the last dose. Male subjects with female partners of childbearing potential must use effective contraception during the trial and for 3 months after the last dose;
11. Subjects must demonstrate good compliance and willingness to participate in follow-up.

Exclusion Criteria:

1. Tumor has significantly invaded adjacent organs (major arteries or trachea) near the esophageal lesion;
2. Presence of supraclavicular lymph node metastasis;
3. Presence of uncontrollable pleural effusion, pericardial effusion, or ascites requiring repeated drainage;
4. Malnutrition with BMI < 18.5 kg/m²; if corrected by symptomatic nutritional support prior to enrollment and approved by the principal investigator, enrollment may still be considered;
5. History of allergy to monoclonal antibodies, any component of adebrelimab, any component of Nimotuzumab, albumin-bound paclitaxel, cisplatin, or other platinum-based drugs;
6. Prior or current treatment with any of the following: (1) Any radiation therapy, chemotherapy, or other anti-neoplastic agents directed at the tumor; (2) Use of immunosuppressive agents or systemic corticosteroids for immunosuppression (dose >10 mg/day prednisone or equivalent) within 2 weeks prior to first study drug administration; Inhaled or topical steroids and corticosteroid replacement therapy at a dose >10 mg/day of prednisone or equivalent are permitted in the absence of active autoimmune disease; (3) Received a live attenuated vaccine within 4 weeks prior to the first dose of study drug; (4) Undergone major surgery or sustained severe trauma within 4 weeks prior to the first dose of study drug;
7. Presence of any active autoimmune disease or history of autoimmune disease, including but not limited to: interstitial pneumonia, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism (may be considered for inclusion after hormone replacement therapy); Individuals with psoriasis or childhood asthma/allergies that have achieved complete remission and require no intervention in adulthood may be considered for inclusion; however, patients requiring medical intervention with bronchodilators are excluded;
8. History of immunodeficiency, including HIV-positive status, or other acquired or congenital immunodeficiency disorders, or history of organ transplantation or allogeneic bone marrow transplantation;
9. Uncontrolled cardiac clinical symptoms or disease, including but not limited to: (1) NYHA Class II or higher heart failure, (2) unstable angina, (3) myocardial infarction within the past year, (4) clinically significant supraventricular or ventricular arrhythmias uncontrolled despite clinical intervention or with poor control after intervention;
10. Severe infection (CTCAE ≥ Grade 2) within 4 weeks prior to first study drug administration, such as severe pneumonia requiring hospitalization, bacteremia, or infection-related complications; exclusion if baseline chest imaging indicates active pulmonary inflammation, or if symptoms/signs of infection or need for oral/IV antibiotics exist within 14 days prior to first study drug administration (excluding prophylactic antibiotic use);
11. Active pulmonary tuberculosis infection identified through medical history or CT examination; history of active pulmonary tuberculosis infection within 1 year prior to enrollment; or history of active pulmonary tuberculosis infection more than 1 year prior without formal treatment;
12. Active hepatitis B (HBV DNA ≥ 2000 IU/mL or 10^4 copies/mL) or hepatitis C (HCV antibody positive with HCV RNA above the lower limit of detection of the assay method);
13. Imaging demonstrating tumor invasion into the perivascular space of a major vessel, or patients judged by the investigator to be at high risk of fatal hemorrhage due to tumor invasion into a major vessel during the study period;
14. Patients diagnosed with other malignancies within 5 years prior to first administration of the study drug, unless the malignancy carries a low risk of metastasis or mortality (5-year survival rate > 90%), such as adequately treated basal cell carcinoma, squamous cell carcinoma of the skin, or cervical carcinoma in situ, which may be considered for inclusion;
15. Patients with uncontrolled hypertension despite antihypertensive therapy (systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100 mmHg); or patients requiring two or more antihypertensive agents to control blood pressure; patients with a history of hypertensive crisis or hypertensive encephalopathy;
16. Pregnant or lactating women;
17. Other factors deemed by the investigator to potentially necessitate premature study discontinuation, such as concomitant treatment for other serious illnesses (including psychiatric disorders), alcohol abuse, substance misuse, or familial/social factors that may compromise subject safety or compliance.
18. Other circumstances deemed unsuitable for inclusion by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
pCR, Pathological Complete Response | From patient enrollment to the end of surgery, assessed up to 12 months

SECONDARY OUTCOMES:
MPR，Main Pathological Response Rate | From patient enrollment to the end of surgery, assessed up to 12 months
Margin-free (R0) resection rate | From patient enrollment to the end of surgery, assessed up to 12 months
EFS, Event free survival | The time from the start of treatment to the first occurrence of any of the following events: disease progression beyond surgical intervention, local or distant recurrence, death from any cause, etc. assessed up to 36 months
OS, Overall Survival | From the start of treatment to death from any cause，assessed up to 60 months
Adverse events rate (CTCAE 5.0) | From the start of enrollment to the completion of the study，assessed up to 60 months
  All treatment-related adverse events, immune-related adverse events, and adverse events of grade 3 or higher, as defined by the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

IPD SHARING:
Plan to Share IPD: No